CLINICAL TRIAL: NCT02718482
Title: Multicentric, Randomized Phase II Trial for the Treatment of Patients With Relapsed Osteosarcoma
Brief Title: Phase II Trial for the Treatment of Relapsed Osteosarcoma
Acronym: OsteoREC2015
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not adequate enrollment (sample size not possible to reach)
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OsteoREC2015
Record Dates: First submitted 2016-03-02; First posted 2016-03-24 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: OSTEOSARCOMA
MeSH Terms: conditions — Osteosarcoma | interventions — Gemcitabine; Docetaxel; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine and Docetaxel (Experimental): Gemcitabine i.v. 900 mg/m2 in 30 min on day 1 and day 8 every 3 weeks Docetaxel i.v. 75 mg/m2 in 60 min on day 8 every 3 weeks
  Interventions: Drug: Gemcitabine and Docetaxel
- Ifosfamide (Experimental): Ifosfamide i.v. 14 g/m2 continous dose for 14 days every 3 weeks
  Interventions: Drug: Ifosfamide

INTERVENTIONS:
Drug: Gemcitabine and Docetaxel — Treatment with gemcitabine and docetaxel at day 1 and day 8 n a 3 weeks cycle
  Arms: Gemcitabine and Docetaxel
Drug: Ifosfamide — Treatment arm with high doses of ifosfamide continous infusion for 14 days in a 3 weeks cycle
  Other Names: High doses ifosfamide
  Arms: Ifosfamide

SUMMARY:
Phase II randomized study for the comparison of the Gemcitabine plus Docetaxel and the Ifosfamide treatment of patients with relapsed osteosarcoma

DETAILED DESCRIPTION:
Patients with relapsed osteosarcoma will be randomized to receive Gemcitabine plus Docetaxel or High Doses Ifosfamide (continuous infusion) every 3 weeks, up to 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high grade osteosarcoma recurrence
* Resectable or unresectable recurrence disease within 24 months from the initial diagnosis
* Pleuro-pulmonary recurrence with more than 2 nodules within 24 months from the initial diagnosis
* Unresectable first relapse within 24 months from the initial diagnosis
* Resectable or unresectable second of further recurrence of high grade osteosarcoma
* Age at diagnosis at least 4years.
* Karnofsky performance status over 60%.
* Renal function and hepatic In normal limits for age.
* L eft ejection ventricular fraction over 50%.
* White blood cells over 3000 million/liter and platelets 100000 million/liter
* Birth potential female must agreed to contraception
* Signed written informed consent

Exclusion Criteria:

* Contraindication to the use of any study drugs
* Mental, social and geographic conditions which fail to ensure adequate adherence to the study
* Hepatitis and human immunodeficiency virus active infection
* Pregnancy or breast-feeding
* Previous treatment with Gemcitabine, Docetaxel and Ifosfamide

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | at 6 months from randomization
  Survival without progression of disease assessed at 6 months from randomization

SECONDARY OUTCOMES:
Overall Response Rate | After 6, 12 and 18 weeks
  Rate of tumor response assessed after cycle 2, 4 and 6
Overall Survival | At patient death or at last available follow-up
  From date of starting therapy until the date of death from any cause, whichever came first, assessed up to 60 months
Post treatment Surgery Rate | After 6, 12 and 18 weeks
  Rate of patients who will require surgery after 2, 4 and 6 study treatment cycles
Adverse Events Incidence | Every 3 weeks up to 22 weeks
  Number and grade of adverse events related to the study treatments
Quality of life assesment: data will be collected by using specific oncologic Quality of Life instruments | After 6, 12 and 18 weeks and at 12 Months after end of treatment
  Quality of Life evaluation related to received chemotherapy
Duration of hospitalization | After 1,3, 4, 6, 7, 9, 10, 12, 13, 15, 16 and 18 weeks
  Number of days spent in hospital related to treatment received

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Ferrari, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (10):
- Italy (10):
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Ospedale Gradenigo, Torino, TO
  - Istituti Ortopedici Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna
  - A.O. Universitaria Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - FONDAZIONE IRCCS Istituto Nazionale dei Tumori, Milan
  - Università seconda di Napoli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Istituto Regina Elena - IFO, Rome
  - Ospedale Infantile Regina Margherita - Unit of Paediatric Oncoematology, Torino

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Saeter G, Hoie J, Stenwig AE, Johansson AK, Hannisdal E, Solheim OP. Systemic relapse of patients with osteogenic sarcoma. Prognostic factors for long term survival. Cancer. 1995 Mar 1;75(5):1084-93. doi: 10.1002/1097-0142(19950301)75:53.0.co;2-f. PMID 7850705
- [Background] Bacci G, Briccoli A, Ferrari S, Ruggieri P, Avella M, Casadei R, Battistini A, Picci P. [Osteosarcoma of the extremities metastatic at presentation. Results obtained with primary chemotherapy followed by simultaneous resection of the primary and metastatic lesion]. Minerva Chir. 1993 Jan;48(1-2):35-45. Italian. PMID 8464555
- [Background] Bielack SS, Kempf-Bielack B, Delling G, Exner GU, Flege S, Helmke K, Kotz R, Salzer-Kuntschik M, Werner M, Winkelmann W, Zoubek A, Jurgens H, Winkler K. Prognostic factors in high-grade osteosarcoma of the extremities or trunk: an analysis of 1,702 patients treated on neoadjuvant cooperative osteosarcoma study group protocols. J Clin Oncol. 2002 Feb 1;20(3):776-90. doi: 10.1200/JCO.2002.20.3.776. PMID 11821461
- [Background] Meazza C, Casanova M, Luksch R, Podda M, Favini F, Cefalo G, Massimino M, Ferrari A. Prolonged 14-day continuous infusion of high-dose ifosfamide with an external portable pump: feasibility and efficacy in refractory pediatric sarcoma. Pediatr Blood Cancer. 2010 Oct;55(4):617-20. doi: 10.1002/pbc.22596. PMID 20589638